CLINICAL TRIAL: NCT05664048
Title: Effects of Dry Heat Application on Menstrual Symptoms and Pain: A Randomized Controlled Trial
Brief Title: Effects of Dry Heat Application for Menstrual Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-045
Record Dates: First submitted 2022-12-10; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Reproductive Health
Keywords: Menstruation; Hot pack application; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry heat application group (Experimental): The participants were informed that they could use the thermophore whenever they felt pain throughout the menstrual cycle. On the first day of the period, they were asked to complete the "Visual Analog Scale" and "Menstrual Symptom Questionnaire" before using the thermophore; apply heat on their sole whenever they felt pain in the first three days of the menstrual period when pain is more intense; rate level of pain twice a day at 12-hour intervals on a daily basis, using the "Visual Analog Scale"; and complete the "Menstrual Symptom Questionnaire" on the last day of the period. On the other hand, the students in the control group completed only the related forms. The students who were previously trained on heat application were trained once again by the researcher as a reminder and then their written consents were obtained through the informed consent form.
  Interventions: Behavioral: Dry heat application
- Control group (No Intervention): The students in the control group completed only the related forms ("Visual Analog Scale" and "Menstrual Symptom Questionnaire") in the period of the menstruation.

INTERVENTIONS:
Behavioral: Dry heat application — Self- dry heat application on the foot during menstrual period with pain.
  Arms: Dry heat application group

SUMMARY:
This randomized controlled trial was to determine the effect of dry heat applied on foot base of the 65 nursing students on menstrual symptoms and pain. A statistically significant difference was found between the three-day Visual Analog Pain Scale in both intervention and control groups. However, there was no difference between Menstruation Symptom Scale subscale and total score avg of the intervention and control groups. Applying hot pack to the sole of the foot can be expressed as an effective method to reduce pain. However, due to premenstrual syndrome is a complex process, the reduction of pain in the later days of the menstrual cycle in both groups can be psychological or be explained for physiological reasons.

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled trial, a non-blinded between 30 September 2019 and 29 November 2019. In the first stage of the present study, the Premenstrual Syndrome Scale was used for all participants and the study was continued with the students with premenstrual syndrome symptoms based on the data acquired from the Premenstrual Syndrome Scale. This stage was used only for restricting the sample group, rather than diagnosing or treating the students. In the second stage, the randomization of students included in the sample group was presented according to the CONSORT diagram. The population of the study consisted of 452 female nursing students studying in the faculty of health sciences in a university. The students (n=75) who were absent in the school, took analgesics during the study, and did not agree to participate in the study, were excluded from the study. The students, who had no diagnosis of psychiatric disorder and history of endometriosis, stated that they menstruated regularly (between 22-35 days), did not use complementary and alternative treatments such as analgesics or massage throughout the study, had no diabetes or neuropathic problem causing nerve injury, did not take oral contraceptives, were over 18 years, and agreed to participate in the study, were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* having no diagnosis of psychiatric disorder and history of endometriosis
* stated that they menstruated regularly (between 22-35 days),
* not use complementary and alternative treatments such as analgesics or massage throughout the study,
* having no diabetes or neuropathic problem causing nerve injury,
* not take oral contraceptives,
* were over 18 years,
* agreed to participate in the study

Exclusion Criteria:

* analgesics during the study
* not agree to participate in the study

Ages: 18 Years to 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 65 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Pain due to menstruation. | 10 days.
  Visual Analog Scale was used.Used for measurement and follow up of level of pain this scale is a simple method. In a 10-cm horizontal scale, '0' indicates no pain and '10' indicates worst pain. The students were asked to rate their level of pain during their last period by giving a score between 0 and 10 points.
Menstrual Symptoms. | 10 days.
  Menstrual Symptom Questionnaire was used.

CONTACTS AND LOCATIONS:
Overall Officials: Kıvan Çevik Kaya, Assoc.Prof., Principal Investigator — Celal Bayar University
Locations (1):
- Dilay Açıl, Yunusemre, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be given if it's necessary and if it is not problem for ethical office.

REFERENCES:
- [Background] Negriff S, Dorn LD, Hillman JB, Huang B. The measurement of menstrual symptoms: factor structure of the menstrual symptom questionnaire in adolescent girls. J Health Psychol. 2009 Oct;14(7):899-908. doi: 10.1177/1359105309340995. PMID 19786516
- [Result] Karout S, Soubra L, Rahme D, Karout L, Khojah HMJ, Itani R. Prevalence, risk factors, and management practices of primary dysmenorrhea among young females. BMC Womens Health. 2021 Nov 8;21(1):392. doi: 10.1186/s12905-021-01532-w. PMID 34749716
- [Result] Jo J, Lee SH. Heat therapy for primary dysmenorrhea: A systematic review and meta-analysis of its effects on pain relief and quality of life. Sci Rep. 2018 Nov 2;8(1):16252. doi: 10.1038/s41598-018-34303-z. PMID 30389956
- [Result] Alsaleem MA. Dysmenorrhea, associated symptoms, and management among students at King Khalid University, Saudi Arabia: An exploratory study. J Family Med Prim Care. 2018 Jul-Aug;7(4):769-774. doi: 10.4103/jfmpc.jfmpc_113_18. PMID 30234051

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT05664048/Prot_SAP_000.pdf